CLINICAL TRIAL: NCT00462722
Title: COX Inhibition & Musculoskeletal Responses to Exercise
Brief Title: Myogenic and Osteogenic Responses to eXercise and Ibuprofen
Acronym: MOXI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: 06-0769; R01AG018857 (NIH)
Record Dates: First submitted 2007-04-17; First posted 2007-04-19 (Estimated); Results first posted 2015-08-10 (Estimated); Last update posted 2015-11-02 (Estimated); Status verified 2015-10

CONDITIONS: Aging; Physical Fitness
Keywords: body composition; bone density; cyclooxygenase inhibitor; bone metabolism; muscle function; muscle strength
MeSH Terms: interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo pre and post exercise (Placebo Comparator): placebo before and after musculoskeletal-loading exercise
  Interventions: Drug: Placebo; Behavioral: musculoskeletal-loading exercise
- Placebo pre and ibuprofen post exercise (Experimental): placebo before and ibuprofen after musculoskeletal-loading exercise
  Interventions: Drug: Ibuprofen; Drug: Placebo; Behavioral: musculoskeletal-loading exercise
- Ibuprofen pre and placebo post exercise (Experimental): ibuprofen before and placebo after musculoskeletal-loading exercise
  Interventions: Drug: Ibuprofen; Drug: Placebo; Behavioral: musculoskeletal-loading exercise

INTERVENTIONS:
Drug: Ibuprofen — 400 mg with each exercise session (up to 5 days per week) for 9 months
  Other Names: Motrin; Advil
  Arms: Ibuprofen pre and placebo post exercise; Placebo pre and ibuprofen post exercise
Drug: Placebo — with each exercise session (up to 5 days per week) for 9 months
Behavioral: musculoskeletal-loading exercise — Exercise training program designed to increase bone and muscle mass, including weight lifting and weight-bearing exercises such as jumping in place and treadmill walking up to 5 days per week for 9 months

SUMMARY:
The purpose of this study is to determine if the use of ibuprofen blocks the benefits of exercise to build bone and muscle mass.

DETAILED DESCRIPTION:
People are advised to engage in weight-bearing physical activity to help prevent the loss of bone and muscle mass that occurs with aging. There is evidence from studies of animals that non-steroidal anti-inflammatory drugs (NSAIDS), such as ibuprofen, block some of the bone- and muscle-building effects of exercise. The aim of this study is to determine whether use of ibuprofen, either before or after exercise, blocks the benefits of exercise training on bone and skeletal muscle in older women and men. The hypothesis is that taking ibuprofen before exercise will block some of the effects of exercise training to increase bone density and muscle mass.

Women and men aged 60-75 years will complete a supervised, 9-month exercise training program designed to increase bone and muscle mass. The training will include weight lifting and weight-bearing exercises, such as jumping in place and treadmill walking, up to 5 days per week. Participants will be randomly assigned to take 1 of 3 study pill combinations before and after each exercise session. The combinations of study pills will be: placebo before/placebo after, placebo before/ibuprofen after, or ibuprofen before/placebo after. The dose of ibuprofen will be 400 mg. Bone density of the hip and spine, body composition (total body muscle and fat), and markers of bone turnover in the blood will be measured before and after 4.5 and 9 months of training. Muscle cross-sectional area of the thigh will be measured by CT before and after 9 months of training. A subset of participants will have biopsies of the thigh muscle before and after training to measure proteins and genes associated with muscle build-up and breakdown.

Volunteers who do not use ibuprofen, aspirin, or acetaminophen more than 3 days per month will be enrolled. People with intolerance to ibuprofen or related drugs, cardiovascular disease, or orthopedic problems that limit exercise will be excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60 to 75 years
* Willing to participate in a 9-month supervised exercise program that will start at a moderate intensity and gradually progress to a vigorous intensity
* Not currently performing regular, moderate-to-vigorous weight-bearing or weight-lifting exercise
* Average use of NSAIDs (including low-dose aspirin) or acetaminophen less than 3 days per month

Exclusion Criteria:

* Relative or absolute contraindications to regular use of NSAIDs
* Known allergy or intolerance (heartburn, stomach pain, nausea, vomiting) to NSAIDs; controlled GERD(Gastroesophageal Reflux Disease), if not related to NSAID use, will not be an exclusion criterion
* Proton Pump Inhibitor (PPI) use if dose is unstable or if using for less than 6 months prior to study enrollment
* History of peptic ulcer or upper GI bleeding
* Anemia
* Asthma with bronchospasm induced by aspirin or other NSAIDs
* Moderate or severe renal impairment defined as a calculated creatinine clearance
* Chronic hepatobiliary disease, conservatively defined as liver function tests greater than 1.5 times the upper limit of normal (if such values are obtained on initial screening and thought to be transient in nature, repeated testing will be allowed)
* Hyperkalemia
* Osteoporosis
* Diabetes mellitus requiring pharmacologic therapy
* Congestive heart failure
* Uncontrolled hypertension; use of thiazide diuretics will be allowed if on a stable dose for at least 6 months
* Cardiovascular disease
* Thyroid dysfunction
* Orthopedic problems (e.g., chronic back pain, severe osteoarthritis, rheumatoid arthritis) that limit the ability to perform vigorous exercise and increase the likelihood that the volunteer will use pain medications other than the study pills
* Certain use of medications, including

  * Drugs that are known to alter bone metabolism (e.g., estrogen, SERMs(Selective estrogen-receptor modulators), testosterone, bisphosphonates, teriparatide, calcitonin, GnRH(Gonadotropin-releasing hormone) agonists)
  * Chronic use of oral corticosteroids or any use in the previous 6 months (use of inhaled steroids will not be an exclusion criterion based on a meta-analysis documenting that the effect on bone is not significant)
  * Average use of acetaminophen or NSAIDs, including low-dose aspirin, greater than 3 days per month; volunteers using aspirin for primary prevention may enroll in the study if they discontinue aspirin therapy for the 9-month intervention period
  * Anticoagulants (e.g., warfarin, clopidogrel)
  * Narcotics

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2007-07; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Kohrt, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Aurora, Colorado, United States

REFERENCES:
- [Background] Chow JW, Chambers TJ. Indomethacin has distinct early and late actions on bone formation induced by mechanical stimulation. Am J Physiol. 1994 Aug;267(2 Pt 1):E287-92. doi: 10.1152/ajpendo.1994.267.2.E287. PMID 8074209
- [Background] Li J, Burr DB, Turner CH. Suppression of prostaglandin synthesis with NS-398 has different effects on endocortical and periosteal bone formation induced by mechanical loading. Calcif Tissue Int. 2002 Apr;70(4):320-9. doi: 10.1007/s00223-001-1025-y. Epub 2002 Mar 26. PMID 12004337
- [Background] Trappe TA, White F, Lambert CP, Cesar D, Hellerstein M, Evans WJ. Effect of ibuprofen and acetaminophen on postexercise muscle protein synthesis. Am J Physiol Endocrinol Metab. 2002 Mar;282(3):E551-6. doi: 10.1152/ajpendo.00352.2001. PMID 11832356
- [Derived] Wherry SJ, Wolfe P, Schwartz RS, Kohrt WM, Jankowski CM. Ibuprofen taken before exercise blunts the IL-6 response in older adults but does not alter bone alkaline phosphatase or c-telopeptide. Eur J Appl Physiol. 2021 Aug;121(8):2187-2192. doi: 10.1007/s00421-021-04691-8. Epub 2021 Apr 19. PMID 33876259

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo Pre and Post Exercise | Ibuprofen Pre and Placebo Post Exercise | Placebo Pre and Ibuprofen Post Exercise
Started | 50 | 55 | 54
Completed | 37 | 51 | 42
Not Completed | 13 | 4 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Pre and Post Exercise | Ibuprofen Pre and Placebo Post Exercise | Placebo Pre and Ibuprofen Post Exercise | Total
Number analyzed (Participants) | 37 | 51 | 42 | 130
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (4) | 64 (4) | 66 (4) | 64 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 32 | 27 | 82
  Male | 14 | 19 | 15 | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 1 | 5
  Not Hispanic or Latino | 35 | 49 | 41 | 125
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1 | 2
  Asian | 1 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 5 | 7
  White | 33 | 47 | 35 | 115
  More than one race | 3 | 0 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 37 | 51 | 42 | 130

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline in Lumbar Spine Bone Mineral Density (BMD) at 9 Months
Time Frame: Baseline and after 9 months of training
Population: One participant in the "Ibuprofen pre and placebo post exercise" group had an uninterpretable spine scan.
Measure: Mean (Standard Deviation); unit: Percentage change in lumbar spine BMD
Arm/Group | Placebo Pre and Post Exercise | Ibuprofen Pre and Placebo Post Exercise | Placebo Pre and Ibuprofen Post Exercise
Number analyzed (Participants) | 37 | 50 | 42
Percentage change in lumbar spine BMD | 1.3 (2.8) | 1.5 (2.5) | 0.9 (2.2)

2. Primary Outcome: Percentage Change From Baseline in Total Hip Bone Mineral Density (BMD) at 9 Months
Time Frame: Baseline and after 9 months of training
Population: One participant in the "Placebo pre and post exercise" group and two participants in the "Ibuprofen pre and placebo post exercise" group had uninterpretable hip scans.
Measure: Mean (Standard Deviation); unit: percentage change in total hip BMD
Arm/Group | Placebo Pre and Post Exercise | Ibuprofen Pre and Placebo Post Exercise | Placebo Pre and Ibuprofen Post Exercise
Number analyzed (Participants) | 36 | 49 | 42
percentage change in total hip BMD | 0.5 (2.6) | 0.0 (1.9) | -0.3 (2.0)

3. Primary Outcome: Change From Baseline in Fat-free Mass at 9 Months
Time Frame: Baseline and after 9 months of training
Measure: Mean (Standard Deviation); unit: change in kg
Arm/Group | Placebo Pre and Post Exercise | Ibuprofen Pre and Placebo Post Exercise | Placebo Pre and Ibuprofen Post Exercise
Number analyzed (Participants) | 37 | 51 | 42
change in kg | 0.6 (1.1) | 0.4 (1.6) | 0.6 (1.4)

4. Secondary Outcome: Percentage Change From Baseline in Femoral Neck Bone Mineral Density (BMD) at 9 Months
Time Frame: Baseline and after 9 months of training
Population: One participant in the "Placebo pre and post exercise" group and two participants in the "Ibuprofen pre and placebo post exercise" group had uninterpretable spine scans.
Measure: Mean (Standard Deviation); unit: percentage change in BMD
Arm/Group | Placebo Pre and Post Exercise | Ibuprofen Pre and Placebo Post Exercise | Placebo Pre and Ibuprofen Post Exercise
Number analyzed (Participants) | 36 | 49 | 42
percentage change in BMD | 0.2 (2.9) | 0.2 (2.8) | -0.1 (2.1)

5. Secondary Outcome: Percentage Change From Baseline in Trochanter Bone Mineral Density (BMD) at 9 Months
Time Frame: Baseline and after 9 months of training
Measure: Mean (Standard Deviation); unit: percentage change in BMD
Arm/Group | Placebo Pre and Post Exercise | Ibuprofen Pre and Placebo Post Exercise | Placebo Pre and Ibuprofen Post Exercise
Number analyzed (Participants) | 36 | 49 | 42
percentage change in BMD | 1.1 (3.1) | 0.0 (2.3) | -0.1 (2.7)

6. Secondary Outcome: Percentage Change From Baseline in Sub-trochanter Bone Mineral Density (BMD) at 9 Months
Time Frame: Baseline and after 9 months of training
Population: One participant in the "Placebo pre and post exercise" group and two participants in the "Ibuprofen pre and placebo post exercise" groups had uninterpretable hip scans.
Measure: Mean (Standard Deviation); unit: percentage change in BMD
Arm/Group | Placebo Pre and Post Exercise | Ibuprofen Pre and Placebo Post Exercise | Placebo Pre and Ibuprofen Post Exercise
Number analyzed (Participants) | 36 | 49 | 42
percentage change in BMD | 0.5 (3.4) | 0.0 (2.3) | -0.3 (2.5)

7. Secondary Outcome: Change in Thigh Cross-sectional Muscle Area
Time Frame: Baseline and after 9 months of training
Population: Because of the costs associated with data analysis for this secondary outcome, we did not pursue the analysis after learning the results of the primary outcome (fat-free mass).
Arm/Group | Placebo Pre and Post Exercise | Ibuprofen Pre and Placebo Post Exercise | Placebo Pre and Ibuprofen Post Exercise
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Bone Turnover Markers
Time Frame: Baseline, and after 4.5 & 9 months of training
Population: Because of the costs associated with the assays and data analysis of bone turnover markers, we did not pursue data collection after learning of the primary outcomes (changes in BMD).
Arm/Group | Placebo Pre and Post Exercise | Ibuprofen Pre and Placebo Post Exercise | Placebo Pre and Ibuprofen Post Exercise
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Expression of Selected Proteins and Genes Associated With Muscle Build-up and Breakdown
Time Frame: Baseline and after 9 months of training
Population: Because of the costs associated with gene and protein expression techniques and data reduction, we did not pursue this secondary outcome after learning the results of the primary outcome (change in fat-free mass).
Arm/Group | Placebo Pre and Post Exercise | Ibuprofen Pre and Placebo Post Exercise | Placebo Pre and Ibuprofen Post Exercise
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Placebo Pre and Post Exercise | Ibuprofen Pre and Placebo Post Exercise | Placebo Pre and Ibuprofen Post Exercise
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/51 | 0/42
Other Adverse Events (participants affected / at risk) | 0/37 | 1/51 | 0/42
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Pre and Post Exercise (N=37) | Ibuprofen Pre and Placebo Post Exercise (N=51) | Placebo Pre and Ibuprofen Post Exercise (N=42)
change in estimated glomerular filtration rate (eGFR) (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) — Decrease in eGFR > 25% triggered discontinuation of study drug

LIMITATIONS AND CAVEATS:
The study did not include a no-exercise control group. The variability in the BMD responses was greater than expected.

The results may be specific to ibuprofen and not to other NSAIDs.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No